CLINICAL TRIAL: NCT03033875
Title: Testing Tele-Savvy, an On-line Psychoeducation Program for Dementia Family Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Kenneth Hepburn, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00092812; 1R01AG054079-01 (NIH)
Record Dates: First submitted 2017-01-25; First posted 2017-01-27 (Estimated); Results first posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Alzheimer Disease; Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 2:2:1 ratio to the Tele-Savvy intervention, Healthy Living intervention, or usual care condition. Participants in the Healthy Living and usual care arms can take part i the Tele-Savvy intervention after a delay of 6 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tele-Savvy Group (Experimental): Informal caregivers of persons living with Alzheimer's disease will be randomized to participate in the Tele-Savvy program immediately.
  Interventions: Behavioral: Tele-Savvy
- Attention Control Group (Other): Informal caregivers of persons living with Alzheimer's disease will be randomized to participate in the Healthy Living Education Program. Persons in this group will be able to participate in the Tele-Savvy intervention after a delay of 6 months.
  Interventions: Behavioral: Healthy Living Education Program
- Usual Care Group (No Intervention): Informal caregivers of persons living with Alzheimer's disease will be randomized to continue to receive care through whatever arrangement has been in place. Persons in this group will be able to participate in the Tele-Savvy intervention after a delay of 6 months.

INTERVENTIONS:
Behavioral: Tele-Savvy — The Tele-Savvy program engages groups of six dementia family caregivers in a program that extends over 43 days. The program begins with a scheduled 75-minute group videoconference led by facilitators; similar group videoconferences then take place weekly for six weeks. In between the video-conferences, caregivers will receive daily emails with links to 5-15 minute on-line video lessons that can be watched on their own schedule as often as they wish. The videoconferences allow caregivers to report enactment of learned and self-developed management strategy behaviors into their own caregiving and allow them to raise questions. Each daily video presents a teaching point linked to the overall curriculum. The lesson is carried forward by brief, scripted talks by experts or is enacted in vignettes in which a fictional family caring for a father living with Alzheimer's demonstrates effective caregiving techniques linked to the day's teaching points.
  Arms: Tele-Savvy Group
Behavioral: Healthy Living Education Program — The Healthy Living Education Program contains video and text materials on exercise, diet, and healthy living. Participants will be asked to log into the Canvas site daily over the course of six weeks to view the videos. Each participant will also receive 7 weekly brief scripted phone or video calls from a project facilitator to inquire about participants' use of the materials. Additionally, all participants will convene weekly for a video conference centered on the application of healthy living strategies. Facilitators will greet and check in with each of the caregivers, coach and debrief caregivers on the homework, answer questions and/or respond to feedback about the week's material, review key points and concepts from the week's video sessions and introduce new material, report on any activities that caregivers may have implemented based on the materials, and provide homework assignments.
  Arms: Attention Control Group

SUMMARY:
The purpose of this study is to test the psychoeducational program "Tele-Savvy." Tele-Savvy is an internet based, group education program developed from an in person program called Savvy Caregiver. Participants will be randomly assigned to either the Tele-Savvy group (receiving only the Tele-Savvy education) or the Healthy Living Education Program (receiving healthy lifestyle education and then Tele-Savvy education 6 months later) or a usual care group (receiving Tele-Savvy education 6 months later). Each program takes 43 days to complete.

DETAILED DESCRIPTION:
This study addresses the reliance on family members to provide virtually all community-based care for 5.3 million persons living with Alzheimer's disease and other dementias, a population that will likely triple in the next 35 years. Unless researchers soon find a way to prevent and cure dementing illnesses like Alzheimer's, the country will continue to face an urgent need to find ways to sustain and bolster the capacity of these family caregivers to manage the multiple daily care challenges they face and to preserve their well-being while doing so. Without family caregivers, the burden of care could well overwhelm the formal components of our care system. A number of psychoeducation programs for caregivers have been effective in relieving distress, increasing self-efficacy, managing caregiving challenges, and enabling caregivers to sustain care over longer periods of time. However, many Alzheimer's caregivers cannot take part in these programs because virtually all such programs require caregivers to arrange care for the care recipient while the caregivers attend the programs. These are obstacles in rural or remote areas where transportation issues further restrict caregivers' already limited access to caregiver programs, but they are no less a problem in inner cities and suburbs. These obstacles highlight a substantial challenge to our ability to rely on caregivers as a continuing care resource for persons living with Alzheimer's disease: there is a need for theory-driven psychoeducation programs that can be made readily available to caregivers who may not be able to attend in-person programs.

This is a randomized trial to test a program designed to meet this critical need. This study will test Tele-Savvy, an internet-based program based on the widely disseminated, in-person Savvy Caregiver psychoeducation program. Delivered in scheduled videoconferences and independently viewed on-line video lessons, Tele-Savvy aims to develop/enhance caregivers' skills and caregiving mastery, reduce adverse effects of caregiving, and improve the quality of the lives of caregivers and care recipients.

Caregivers will be randomly assigned either to immediate Tele-Savvy participation groups or to attention control or usual care groups that are invited to participate in Tele-Savvy six months after baseline data collection. Each program takes 43 days to complete. In those 43 days, participants will be asked to take part in a video conference once per week (60-90 minutes) and view daily video lessons (7-15 minutes). The study includes 5 interviews over the course of the 12 month study; the interviews at baseline and months 3 and 6 assess the study outcome measures. These interviews will discuss participant's experience as a caregiver. All interviews will be limited to 60 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Informal caregivers (family/friends) of persons living with Alzheimer's disease or another dementia
* Participants must be providing at least 4 hours per day unpaid assistance, on average, for a person in the early-middle stage of illness (Clinical Dementia Rating of greater than or equal to 1 by home ADC) who is community-dwelling and for whom there is no established plan for institutionalization in the next six months
* Caregiver may or may not reside with their care recipient, but care recipients must live in the community and not in an assisted living facility, nursing home, or another institutional setting
* Must have access to a computer or a mobile device with adequate internet connection, microphone, and speakers (to be able to participate in teleconferences) and be able to use email
* Able to read, speak and understand English

Exclusion Criteria:

* The participant must not be involved in another caregiver training study and must not have participated in in-person Savvy Caregiver Program or Tele-Savvy previously
* Uncorrectable vision or hearing deficits that might impede participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2020-12-04 (Actual); Study Completion 2020-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Hepburn, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

REFERENCES:
- [Background] Kovaleva M, Blevins L, Griffiths PC, Hepburn K. An Online Program for Caregivers of Persons Living With Dementia: Lessons Learned. J Appl Gerontol. 2019 Feb;38(2):159-182. doi: 10.1177/0733464817705958. Epub 2017 May 1. PMID 28460557
- [Background] Kovaleva MA, Bilsborough E, Griffiths PC, Nocera J, Higgins M, Epps F, Kilgore K, Lindauer A, Morhardt D, Shah RC, Hepburn K. Testing Tele-Savvy: Protocol for a randomized controlled trial. Res Nurs Health. 2018 Apr;41(2):107-120. doi: 10.1002/nur.21859. Epub 2018 Feb 5. PMID 29399825
- [Result] Hepburn K, Nocera J, Higgins M, Epps F, Brewster GS, Lindauer A, Morhardt D, Shah R, Bonds K, Nash R, Griffiths PC. Results of a Randomized Trial Testing the Efficacy of Tele-Savvy, an Online Synchronous/Asynchronous Psychoeducation Program for Family Caregivers of Persons Living with Dementia. Gerontologist. 2022 Apr 20;62(4):616-628. doi: 10.1093/geront/gnab029. PMID 33640979
- [Derived] Bonds Johnson K, Higgins M, Epps F, Brewster GS, Alexander K, Hepburn K. Tele-Savvy Outcomes of Non-Hispanic Black American and White Caregivers. Gerontologist. 2024 Jan 1;64(1):gnad044. doi: 10.1093/geront/gnad044. PMID 37067896

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant enrollment began May 18, 2017 and all study follow up was completed by December 4, 2020. Data collection to assess the outcome measures for this study occurred through the interview at month 6. Study activities continued through month 12 while participants in the Attention Control and Usual Care groups had the opportunity to have the Tele-Savvy intervention.
Groups:
- Tele-Savvy Group: Informal caregivers of persons living with Alzheimer's disease randomized to participate in the Tele-Savvy program immediately.
  The Tele-Savvy program engages groups of six dementia family caregivers in a program that extends over 43 days. The program begins with a scheduled 75-minute group videoconference led by facilitators; similar group videoconferences then take place weekly for six weeks. In between the video-conferences, caregivers receive daily emails with links to 5-15 minute on-line video lessons that can be watched on their own schedule as often as they wish. The videoconferences allow caregivers to report enactment of learned and self-developed management strategy behaviors into their own caregiving and allow them to raise questions. Each daily video presents a teaching point linked to the overall curriculum. The lesson is carried forward by brief, scripted talks by experts or is enacted in vignettes in which a fictional family caring for a father living with Alzheimer's demonstrates effective caregiving techniques linked to the day's teaching points.
- Attention Control Group: Informal caregivers of persons living with Alzheimer's disease randomized to participate in the Healthy Living Education Program. Persons in this group were able to participate in the Tele-Savvy intervention after a delay of 6 months.
  The Healthy Living Education Program contains video and text materials on exercise, diet, and healthy living. Participants are asked to log into the Canvas site daily over the course of six weeks to view the videos. Each participant also receives 7 weekly brief scripted phone or video calls from a project facilitator to inquire about participants' use of the materials. Additionally, all participants convene weekly for a video conference centered on the application of healthy living strategies. Facilitators greet and check in with each of the caregivers, coach and debrief caregivers on the homework, answer questions and/or respond to feedback about the week's material, review key points and concepts from the week's video sessions and introduce new material, report on any activities that caregivers may have implemented based on the materials, and provide homework assignments.
- Usual Care Group: Informal caregivers of persons living with Alzheimer's disease randomized to continue to receive care through whatever arrangement has been in place. Persons in this group were able to participate in the Tele-Savvy intervention after a delay of 6 months.
Period: Overall Study
Arm/Group | Tele-Savvy Group | Attention Control Group | Usual Care Group
Started | 96 | 111 | 54
Completed Month 3 Assessment | 71 | 83 | 43
Completed Month 6 Assessment | 73 | 81 | 46
Completed | 77 | 87 | 42
Not Completed | 19 | 24 | 12
Not completed — Withdrawal by Subject | 5 | 9 | 4
Not completed — Other | 14 | 15 | 8

BASELINE CHARACTERISTICS:
Groups:
- Tele-Savvy Group: Informal caregivers of persons living with Alzheimer's disease randomized to participate in the Tele-Savvy program immediately.
- Attention Control Group: Informal caregivers of persons living with Alzheimer's disease randomized to participate in the Healthy Living Education Program. Persons in this group were able to participate in the Tele-Savvy intervention after a delay of 6 months.
- Total: Total of all reporting groups
Arm/Group | Tele-Savvy Group | Attention Control Group | Usual Care Group | Total
Number analyzed (Participants) | 96 | 111 | 54 | 261
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.0 (10.9) | 63.8 (11.6) | 63.7 (10.7) | 64.6 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 73 | 39 | 184
  Male | 24 | 38 | 15 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 92 | 104 | 54 | 250
  Unknown or Not Reported | 4 | 7 | 0 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caregiver race: White | 78 | 75 | 39 | 192
  Caregiver race: African American/Black | 15 | 27 | 15 | 57
  Caregiver race: Asian | 1 | 3 | 0 | 4
  Caregiver race: No answer | 0 | 1 | 0 | 1
  Caregiver race: Other | 2 | 5 | 0 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 96 | 111 | 54 | 261
Age of person cared for [Mean (Standard Deviation); unit: years] | 75.1 (8.6) | 74.4 (10.6) | 74.4 (10.3) | 74.6 (9.8)
Relation to person cared for [Count of Participants; unit: Participants]
  Spouse | 69 | 68 | 35 | 172
  Non-spouse | 27 | 43 | 19 | 89

OUTCOME MEASURES:

1. Primary Outcome: Zarit Burden Inventory (ZBI) Score
Description: The ZBI is a 22 item scale. Each item on the interview is a statement which the caregiver is asked to endorse using a 5-point scale. Response options range from 0 (Never) to 4 (Nearly Always). Total scores range from 0 (low burden) to 88 (high burden)
Time Frame: Baseline, Month 3, Month 6
Population: This analysis includes participants completing the indicated study visit, who also had valid data for this assessment. Some questionnaires had missing or skipped items resulting in removing those participants from the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tele-Savvy Group | Attention Control Group | Usual Care Group
Number analyzed (Participants) | 96 | 111 | 54
score on a scale
  Baseline | 37.34 (13.77) | 35.78 (14.66) | 35.94 (15.99)
  Month 3: number analyzed (Participants) | 69 | 83 | 43
  Month 3 | 35.26 (13.03) | 36.28 (13.49) | 37.82 (15.80)
  Month 6: number analyzed (Participants) | 72 | 80 | 45
  Month 6 | 35.54 (13.63) | 35.91 (12.96) | 37.48 (17.31)

2. Primary Outcome: State-Trait Anxiety Inventory (STAI) State Score
Description: The STAI State (STAI-S) is a 20-item 4-point Likert scale commonly used measure of state anxiety. Respondents report the intensity of their anxiety at that moment on a 4-point scale where 1 = not at all and 4 = very much so. Total scores range from 20 to 80 and higher scores indicate greater anxiety.
Time Frame: Baseline, Month 3, Month 6
Population: This analysis includes participants completing the indicated study visit, who also had valid data for this assessment. One questionnaire had missing or skipped items resulting in one participant being removed from the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tele-Savvy Group | Attention Control Group | Usual Care Group
Number analyzed (Participants) | 96 | 111 | 54
score on a scale
  Baseline | 35.07 (11.96) | 34.61 (13.13) | 33.41 (11.61)
  Month 3: number analyzed (Participants) | 71 | 83 | 43
  Month 3 | 32.90 (12.31) | 32.96 (11.50) | 35.00 (12.15)
  Month 6: number analyzed (Participants) | 72 | 81 | 46
  Month 6 | 31.22 (9.97) | 34.07 (11.83) | 35.41 (12.93)

3. Primary Outcome: Center for Epidemiological Studies Depression Scale - Revised (CESD-R) Score
Description: The CESD-R is a 20 item Likert scale scored 0-3 with somatic and psychological subscales. Total scores range from 0 to 60, with high scores indicating greater depressive symptoms.
Time Frame: Baseline, Month 3, Month 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tele-Savvy Group | Attention Control Group | Usual Care Group
Number analyzed (Participants) | 96 | 111 | 54
score on a scale
  Baseline | 13.14 (9.98) | 12.06 (10.09) | 11.08 (8.25)
  Month 3: number analyzed (Participants) | 71 | 83 | 43
  Month 3 | 10.45 (9.23) | 10.52 (9.18) | 12.07 (8.60)
  Month 6: number analyzed (Participants) | 72 | 81 | 46
  Month 6 | 10.51 (8.16) | 11.65 (10.08) | 12.93 (9.28)

4. Secondary Outcome: Revised Memory and Behavior Problem Checklist (RMBPC) Reaction Score
Description: The RMBPC is a 24-item instrument that assesses behaviors in persons with dementia and caregiver responses to them. Caregiver reactions to behaviors are scored as 0 = not at all upsetting to 4 = extremely upsetting. Total caregiver reaction scores range from 0 to 96 with higher scores indicating greater feelings of being upset by behaviors of those with dementia that they are providing care for.
Time Frame: Baseline, Month 3, Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tele-Savvy Group | Attention Control Group | Usual Care Group
Number analyzed (Participants) | 96 | 110 | 53
score on a scale
  Baseline | 13.84 (9.78) | 12.34 (11.89) | 13.47 (12.30)
  Month 3: number analyzed (Participants) | 70 | 79 | 42
  Month 3 | 10.36 (7.90) | 11.60 (9.01) | 14.50 (10.33)
  Month 6: number analyzed (Participants) | 70 | 78 | 43
  Month 6 | 11.30 (8.26) | 12.28 (9.82) | 15.00 (12.96)

5. Secondary Outcome: Pearlin Mastery, Loss, and Competence - Caregiving Competence Subscale Score
Description: The Caregiving Competence Subscale of the Pearlin Mastery, Loss, and Competence instrument has 4 items that are responded to on a 4-point Likert scale where 1 = not at all and 4 = very much. Total scores for this subscale range from 4 to 16 and higher scores indicate greater feelings of competence with caregiving.
Time Frame: Baseline, Month 3, Month 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tele-Savvy Group | Attention Control Group | Usual Care Group
Number analyzed (Participants) | 96 | 111 | 54
score on a scale
  Baseline | 12.11 (2.12) | 12.44 (1.94) | 12.31 (2.14)
  Month 3: number analyzed (Participants) | 71 | 83 | 43
  Month 3 | 13.21 (1.46) | 12.49 (1.98) | 11.98 (2.27)
  Month 6: number analyzed (Participants) | 72 | 81 | 46
  Month 6 | 13.07 (1.71) | 12.62 (2.15) | 12.52 (2.19)

6. Secondary Outcome: Pearlin Mastery, Loss, and Competence - Management of Situation Subscale Score
Description: The Management of Situation Subscale of the Pearlin Mastery, Loss, and Competence instrument has 4 items that are responded to on a 4-point Likert scale where 1 = never and 4 = very often. Total scores for this subscale range from 4 to 16 and higher scores indicate greater management of caregiving situations.
Time Frame: Baseline, Month 3, Month 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tele-Savvy Group | Attention Control Group | Usual Care Group
Number analyzed (Participants) | 96 | 111 | 54
score on a scale
  Baseline | 11.27 (2.12) | 11.63 (2.00) | 11.43 (1.93)
  Month 3: number analyzed (Participants) | 71 | 83 | 43
  Month 3 | 12.03 (2.06) | 11.35 (2.39) | 11.40 (1.56)
  Month 6: number analyzed (Participants) | 72 | 81 | 46
  Month 6 | 11.93 (2.21) | 11.78 (1.94) | 11.22 (1.59)

7. Secondary Outcome: Perceived Stress Scale (PSS) Score
Description: The PSS is 14-item Likert-type questionnaire. Responses are given on a 5-point scale where 0 = never and 4 = very often. Total scores range from 0 to 56 and certain items are reverse scored so that higher total scores reflect higher perceived stress.
Time Frame: Baseline, Month 3, Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tele-Savvy Group | Attention Control Group | Usual Care Group
Number analyzed (Participants) | 96 | 111 | 54
score on a scale
  Baseline | 23.50 (8.93) | 22.66 (8.21) | 21.73 (7.71)
  Month 3: number analyzed (Participants) | 71 | 83 | 43
  Month 3 | 20.77 (6.93) | 21.24 (7.63) | 23.86 (6.74)
  Month 6: number analyzed (Participants) | 72 | 80 | 46
  Month 6 | 20.72 (7.10) | 22.14 (8.08) | 23.50 (7.36)

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning when individuals gave consent to participate in the study through the final study assessment (up to 12 months).
Arm/Group | Tele-Savvy Group | Attention Control Group | Usual Care Group
All-Cause Mortality (participants affected / at risk) | 0/96 | 0/111 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/96 | 0/111 | 0/54
Other Adverse Events (participants affected / at risk) | 0/96 | 0/111 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-09): https://cdn.clinicaltrials.gov/large-docs/75/NCT03033875/Prot_SAP_001.pdf
  • Informed Consent Form (2019-12-19): https://cdn.clinicaltrials.gov/large-docs/75/NCT03033875/ICF_000.pdf